CLINICAL TRIAL: NCT05263635
Title: Music Therapy in the Treatment of Perioperative Anxiety and Pain-A Randomized, Prospective, Clinical Trial
Brief Title: Music Therapy in the Treatment of Perioperative Anxiety and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Shadyside Hospital Foundation (Other)
Responsible Party: Principal Investigator, Shiv Goel, Chief Anesthesiologist, Principle Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21110130
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Pain, Post Operative; Anxiety; Opioid Use
Keywords: Post operative pain management; music therapy; Post-surgical quality of life; hernia repair surgery; ambulatory breast surgery; cholecystectomy
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Randomized single-blind, comparator controlled trial involving patients undergoing ambulatory breast surgery, laparoscopic cholecystectomy surgery, or laparoscopic hernia repair surgery that score ≥19 on the PROMIS Emotional Distress - Anxiety - Short Form 8a
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy + Standard of Care Enhanced Recovery After Surgery (ERAS) (Experimental): All participants will have complete Enhanced Recovery After Surgery (ERAS) standard of care. A preoperative music intervention will be played first in the preoperative holding area, a second music intervention played immediately following the induction of anesthesia in the operating room, and a third music intervention played in the recovery room when the patient is awake and responsive.
  Interventions: Other: Music therapy; Other: Standard of Care Enhanced Recovery After Surgery (ERAS)
- Standard of Care Enhanced Recovery After Surgery (ERAS) (Active Comparator): Participants randomized into the control group will receive complete Enhanced Recovery After Surgery (ERAS) standard of care and no music therapy sessions.
  Interventions: Other: Standard of Care Enhanced Recovery After Surgery (ERAS)

INTERVENTIONS:
Other: Music therapy — Music therapy will include music intervention based on recommendations from literature such as slow, flowing rhythm, approximately 60-80 beats/minute and played by string instruments, played with a volume of approximately 45 decibel and will be reviewed by qualified music therapists.
  Arms: Music therapy + Standard of Care Enhanced Recovery After Surgery (ERAS)
Other: Standard of Care Enhanced Recovery After Surgery (ERAS) — Patients will receive the standard of care treatment for surgery and post-operative pain management, following the Enhanced Recovery After Surgery (ERAS) protocol

SUMMARY:
A large number of adults who undergo surgery experience perioperative anxiety and pain. The current recommended approach to perioperative pain management is a multimodal approach including opioids. Evidence has demonstrated that the pharmacological management of pain and anxiety is often associated with side effects which limits patient satisfaction and their ability to be discharged from the hospital. Furthermore, it is established that perioperative level of pain is directly correlated to anxiety, depression, and catastrophizing and these are significant predictors for the level of postoperative pain, as well as at the hospital length of stay. Therefore, considerations have been given to the use of non-pharmaceutical complementary approaches to management of anxiety including pre and postoperative use of music. The benefits of music therapy on anxiety has been reported using several surgical models and conditions in adults (cancer, hysterectomy in cancer) and children, prior to surgery and after. The objective of this study is to investigate the effects of music interventions on anxiety and pain in adult populations undergoing diverse types of minor surgery indicate that music therapy significantly reduces both post operative anxiety and pain in adults receiving music interventions before, during, or after surgery.

DETAILED DESCRIPTION:
Screening procedures: There are no specific screening tests or procedures for this research study. Medical records will be examined by an investigator anesthesiologist to determine your eligibility for the study. Eligible subjects will be adults between the ages of 18-70 that also meet the American Society of Anesthesiologists (ASA) physical status I, II, or III, and will be admitted for a scheduled same-day surgery under general anesthesia with a single nerve block including ambulatory breast surgeries, laparoscopic cholecystectomy, and/or laparoscopic hernia repair surgeries. This information will be obtained via medical record.

Enrollment procedures: If a subject qualifies to participate in this study, they will discuss this study with the surgeon investigator and the research study team. They will sign an informed consent form and be enrolled if they choose to participate. They will be asked to complete several questionnaires regarding the subject's baseline anxiety and pain prior to their scheduled surgery. These questionnaires will include the PROMIS Emotional Distress - Anxiety - Short Form 8a, PROMIS Emotional Distress - Depression - Short Form, and the Pain Catastrophizing Scale (PCS).

If the subject remains eligible after their self-report baseline questionnaires, they will be randomized to either the control or intervention group. The control group will receive standard of care treatment during their scheduled surgery but will not be exposed to any music therapy intervention during their hospital stay.

For those assigned to the music therapy group, a preoperative music intervention will be played first in the preoperative area, a second music intervention played immediately following the induction of anesthesia in the operating room, and a third music intervention played in the recovery room when the patient is awake and responsive. The music playing device will be removed after each session.

Music therapy will include music intervention based on recommendations from literature such as slow, flowing rhythm, approximately 60-80 beats/minute and played by string instruments, played with a volume of approximately 45 decibel and will be reviewed by qualified music therapists. Aside from the addition of music intervention, standard of care will not be affected.

Randomization will be completed by a computer-generated, blocked randomization list with equal allocation ratio. After obtaining written informed consent, participants will be subsequently allocated using opaque envelopes to the preoperative music intervention group (music administered during the pre-, intra-, and postoperative period) or the control group.

Regardless of which group a subject is randomized to, participants will expected to complete follow-up questionnaires, including a satisfaction survey at the time of discharge.

Follow-up procedures: Subjects will be contacted via email (REDCap Survey) once daily for 5 days post-op and will be asked to complete the same questionnaires they did at the screening visit. In addition to this, they will also be asked to report a daily pain diary, opioid consumption, and treatment satisfaction also in REDCap Survey.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-70, meeting the American Society of Anesthesiologists (ASA) physical status I, II, or III
* Admitted for a scheduled same-day surgery under general anesthesia with a single nerve block, including ambulatory breast surgery, laparoscopic cholecystectomy or laparoscopic hernia repair surgery

Exclusion Criteria:

* Music other than the intervention planned in the operating room
* ASA status IV
* Planned spinal anesthesia
* Major psychosocial disorders
* Persistent opioid use
* History of drug abuse or alcoholism
* Baseline PROMIS Anxiety score of less than 19 or greater than 35
* Subject is already receiving an alternative intervention for anxiety or pain (i.e aromatherapy, hypnosis, etc)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of music therapy on reducing post-operative opioid requirement | Day of surgery up to 5 days post-operative
  The primary endpoint will be to observe the change in opioid requirement in patients undergoing surgery using the current multimodal Enhanced Recovery After Surgery (ERAS) protocol. This is reported in the consumption of oral morphine mg equivalents (OME).

SECONDARY OUTCOMES:
Pre-operative emotional distress related to anxiety | Baseline, pre-surgery
  Pre-operative emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress -Anxiety- Short Form 8a questionnaire prior to surgery. There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Post-operative change in emotional distress related to anxiety | Day 1, 2, 3, 4, and 5 post-operative
  Post-operative emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress -Anxiety- Short Form 8a questionnaire.There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Pre-operative emotional distress related to depression | Baseline, pre-surgery
  Pre-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form questionnaire prior to surgery. There are 8 questions about how the participant may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Post-operative change in emotional distress related to depression | Day 1, 2, 3, 4, and 5 post-operative
  Pre-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form questionnaire prior to surgery. There are 8 questions about how the participant may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Pre-operative pain rating using the Pain Catastrophizing Scale | Baseline, pre-surgery
  Pre-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome
Post-operative pain rating using the Pain Catastrophizing Scale | Day 1, 2, 3, 4, and 5 post-operative
  Pre-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome.
Length of hospital stay | Day of surgery up to 5 days post-operative
  Evaluate time to hospital discharge from out of OR time in minutes
Incidence of post-operative nausea and vomiting (PONV) | Day of surgery through 5 days post-operative
  Evaluate the number of post-operative nausea and vomiting episodes following surgery.
Post-operative patient satisfaction | Day 5 post-operative
  Participants are asked to assess their overall satisfaction with care upon discharge on a 10-point satisfaction scale of 0 (least satisfaction) to 10 (highest satisfaction). The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a better outcome.
Change in post-operative pain using a numerical rating scale | Day of surgery up to 5 days post-operative
  Numerical Rating Scale (NRS) Pain scores on a scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. higher scores represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Goel, MD, PhD, MBA, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No